CLINICAL TRIAL: NCT00001765
Title: Low Intensity Preparative Regimen Followed by HLA-Matched, Mobilized Peripheral Blood Stem Cell Transplantation for Chronic Granulomatous Disease
Brief Title: Stem Cell Transplant Following Low-Intensity Chemotherapy to Treat Chronic Granulomatous Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980104; 98-I-0104
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-02

CONDITIONS: Chronic Granulomatous Disease
Keywords: Engraftment; Minitransplant; Fludarabine; Neutrophil; Allogenic; Donor Apheresis; Anti-Thymocyte Globin; Cyclophosphamide; Nonmyeloablative Bone Marrow Transplantation; Graft-versus-host Disease; Chronic Granulomatous Disease
MeSH Terms: conditions — Granulomatous Disease, Chronic; Graft vs Host Disease

INTERVENTIONS:
Device: Nexell Isolex with T-cell Depletion
Device: Baxter isolex 300i

SUMMARY:
This study will investigate the safety and effectiveness of a modified stem cell transplant procedure for treating chronic granulomatous disease (CGD) in patients with active infection. CGD is an inherited disorder of neutrophils-a type of infection-fighting white blood cell-that leaves patients vulnerable to life-threatening infections. Transplantation of donated stem cells (cells produced by the bone marrow that mature into the different blood components-white cells, red cells and platelets) can cure CGD. However, this procedure carries a significant risk of death, particularly in patients with active infection, because it requires completely suppressing the immune system with high-dose chemotherapy and radiation. In addition, lymphocytes-another type of infection-fighting white blood cell-from the donor may cause what is called graft vs. host disease (GvHD), in which the donor cells recognize the patient's cells as foreign and mount an immune response to destroy them. To try to reduce these risks, patients in this study will be given low-dose chemotherapy and no radiation, a regimen that is easier for the body to tolerate and involves a shorter period of complete immune suppression. Also, the donor's lymphocytes will be removed from the rest of the stem cells to be transplanted, reducing the risk of GvHD.

Patients with CGD between the ages of age 1 and 55 years old who do not have an active infection and who have a family member that is a well matched donor may be eligible for this study. Candidates will have a medical history, physical examination and blood tests, lung and heart function tests, X-rays of the chest and sinuses, and dental and eye examinations. A bone marrow sample may be taken to evaluate disease status. This test, done under a local anesthetic, uses a special needle to draw bone marrow from the hipbone.

Stem cells will be collected from both the patient and donor. To do this, the hormone G-CSF will be injected under the skin for several days to increase stem cell production. Then, the stem cells will be collected by apheresis. In this procedure the blood is drawn through a needle placed in one arm, pumped into a machine where the desired cells are separated out and removed, and then the rest of the blood is returned through a needle in the other arm.

A large plastic tube (central venous line) is placed into a major vein. It can stay in the body and be used the entire treatment period to deliver the donated stem cells, give chemotherapy or other medications, including antibiotics and blood transfusions, if needed, and withdraw blood samples. Several days before the transplant procedure, patients will start low-dose chemotherapy with cyclophosphamide and fludarabine, two commonly used anti-cancer drugs. They will also be given anti-thymocyte globulin to prevent rejection of the donated cells. When this conditioning therapy is completed, the stem cells will be infused through the central line. Patients will be given cyclosporine by mouth or by vein from 4 days before until 3 months after the stem cell transplant to help prevent rejection.

The average hospital stay for stem cell transplant is 30 days. After discharge, patients will return for follow-up clinic visits weekly or twice weekly for 4 months. These visits will include a symptom check, physical examination, and blood tests. Blood transfusions will be given if needed. Subsequent visits will be scheduled at 4, 6, 12, 18, 24, 30 and 36 months after the transplant or more often if required, and then yearly.

DETAILED DESCRIPTION:
Chronic Granulomatous Disease (CGD) is an inherited disorder of neutrophil function. Patients are profoundly immunocompromised, and are plagued early in life with recurrent, and life threatening infections. Allogeneic stem cell transplantation is the only cure for CGD.

The goal of this phase I/II study is to investigate the safety and efficacy of a novel approach to allogeneic stem cell transplantation aimed at decreasing transplant related morbidity and mortality. We will treat patients with CGD with an allogeneic, G-CSF mobilized peripheral blood stem cell transplant from an HLA identical family member. The graft will be T-cell depleted which will decrease the incidence of acute graft vs. host disease. Donor T-cells will be infused post-transplant if engraftment of donor stem cells is unsatisfactory. The preparative regimen utilized will provide intense immunosuppression without myeloablation. It is designed to allow donor stem cell engraftment while minimizing serious transplant related toxicity.

The end points of this study are engraftment, degree of donor-host chimerism, incidence of acute and chronic GVHD, transplant related morbidity and mortality as well as overall survival.

ELIGIBILITY:
INCLUSION CRITERIA:

PATIENT CRITERIA:

Ages 1 to 55 years

DHR proven Chronic Granulomatous Disease: Includes gp91phox, p47phox, p22phox and p67phox deficiency.

Free of active infection.

Patient has experienced 2 or more prior infections requiring treatment with intravenous anti-bacterial or anti-fungal therapy.

HIV negative.

No major organ dysfunction precluding transplantation.

HLA identical sibling or parent compatible at all 6 of the HLA A, B, and DR antigens by serotyping or DNA typing techniques.

Left ventricular ejection fraction: greater than 40% predicted.

ECOG performance status of 0 or 1.

DONOR CRITERIA:

HLA identical sibling donor or parent donor.

Fit to receive G-CSF and give peripheral blood stem cells (normal blood count, normotensive, no history of stroke, no history of severe heart disease).

Female x-linked CGD carriers must have greater than 30% normal neutrophils.

EXCLUSION CRITERIA:

Patient or donor pregnant.

Age greater than 55 years.

ECOG performance status of 2 or more.

Evidence of rapid deterioration due to progressive infection and/or organ damage.

Left ventricular ejection fraction: greater than or equal to 35 percent predicted.

Creatinine Clearance greater than or equal to 50.

Serum bilirubin greater than or equal to 4 mg/dl, transaminases greater than or equal to 3x upper limit or normal.

HIV negative. Donors who are positive for HBV, HCV or HTLV will be used at the discretion of the investigator.

Malignant diseases liable to relapse or progress within 5 years.

Donors unfit to receive G-CSF and undergo apheresis. (Uncontrolled hypertension, history of stroke, history of heart disease, thrombocytopenia.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1998-04; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ho CM, Vowels MR, Lockwood L, Ziegler JB. Successful bone marrow transplantation in a child with X-linked chronic granulomatous disease. Bone Marrow Transplant. 1996 Jul;18(1):213-5. PMID 8832019
- [Background] Giralt S, Estey E, Albitar M, van Besien K, Rondon G, Anderlini P, O'Brien S, Khouri I, Gajewski J, Mehra R, Claxton D, Andersson B, Beran M, Przepiorka D, Koller C, Kornblau S, Korbling M, Keating M, Kantarjian H, Champlin R. Engraftment of allogeneic hematopoietic progenitor cells with purine analog-containing chemotherapy: harnessing graft-versus-leukemia without myeloablative therapy. Blood. 1997 Jun 15;89(12):4531-6. PMID 9192777
- [Background] Slavin S, Nagler A, Naparstek E, Kapelushnik Y, Aker M, Cividalli G, Varadi G, Kirschbaum M, Ackerstein A, Samuel S, Amar A, Brautbar C, Ben-Tal O, Eldor A, Or R. Nonmyeloablative stem cell transplantation and cell therapy as an alternative to conventional bone marrow transplantation with lethal cytoreduction for the treatment of malignant and nonmalignant hematologic diseases. Blood. 1998 Feb 1;91(3):756-63. PMID 9446633